CLINICAL TRIAL: NCT07108725
Title: The Role of Non-invasive Diffusion-weighted Imaging With MRCP in the Diagnosis of Neoplastic Biliary Obstruction
Brief Title: Non-invasive Diffusion-weighted Imaging With MRCP in the Diagnosis of Neoplastic Biliary Obstruction
Status: Recruiting | Type: Observational
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Hekmat Samir Baumey, Lecturer of Diagnostic Radiology, Damnhour National Medical Institute, The General Authority for Teaching Hospitals and Institutes
Other Study IDs: HMH00013
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Non-invasive Diffusion-weighted Imaging; Magnetic Resonance Cholangiopancreatography; Diagnosis; Neoplastic Biliary Obstruction
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients who are scheduled for magnetic resonance cholangiopancreatography and have undergone conventional imaging
  Interventions: Other: Magnetic Resonance Cholangiopancreatography

INTERVENTIONS:
Other: Magnetic Resonance Cholangiopancreatography — Patients who are scheduled for magnetic resonance cholangiopancreatography and have undergone conventional imaging

SUMMARY:
This study aims to evaluate the diagnostic value of non-invasive diffusion-weighted magnetic resonance imaging (DW-MRI) in detecting neoplastic biliary obstruction.

DETAILED DESCRIPTION:
Both surgeons and endoscopists value accurate approaches for identifying the source of biliary stricture in patients with obstructive jaundice. Cholangiocarcinoma or a benign stricture may cause a biliary stricture. Many imaging methods were used to diagnose the cause of biliary stricture.

Diffusion-weighted magnetic resonance imaging (DW-MRI) has emerged as a non-invasive imaging modality that can potentially differentiate between malignant and benign biliary obstructions based on the measurement of water diffusion in tissues.

The gold standard of the research is endoscopic retrograde cholangiopancreatography (ERCP) and histology. Patients' diagnoses and follow-up were further verified by ERCP or histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with clinically suspected biliary obstruction (e.g., jaundice, elevated liver enzymes, cholestasis).
* Patients who are scheduled for magnetic resonance cholangiopancreatography (MRCP) and have undergone conventional imaging [ultrasound or computed tomography (CT)].
* Patients who will undergo further invasive procedures, e.g., endoscopic retrograde cholangiopancreatography (ERCP), biopsy.

Exclusion Criteria:

* Patients with contraindications to magnetic resonance imaging (MRI) (e.g., pacemakers, metal implants).
* Patients who have previously undergone major biliary surgery or stent placement.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational, diagnostic accuracy study. The study will include patients with suspected biliary obstruction, referred to our hospital for diagnostic imaging.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of magnetic resonance cholangiopancreatography | Immediately after magnetic resonance cholangiopancreatography (Up to 1 hour)
  Sensitivity of magnetic resonance cholangiopancreatography to predict of a tumor will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.